CLINICAL TRIAL: NCT03150030
Title: Hypoglycaemia and Cardiac Arrhythmias in Type 2 Diabetes
Acronym: HYPO-HEART
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Andreas Andersen, MD, PhD-student, University Hospital, Gentofte, Copenhagen
Other Study IDs: H-16046212
Record Dates: First submitted 2017-04-25; First posted 2017-05-11 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2; Arrhythmia, Cardiac
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Arrhythmias, Cardiac | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with type 2 diabetes: Insulin-treated type 2 diabetes with diabetic complications
  Interventions: Other: Combined hyper- and hypoglycaemic clamp; Device: Loop recorder (Reveal LINQ, Medtronic, Minneapolis, MN, USA); Device: Continuous glucose monitoring (iPro2, Medtronic, Minneapolis, MN, USA)
- Healthy controls: Healthy control subjects
  Interventions: Other: Combined hyper- and hypoglycaemic clamp

INTERVENTIONS:
Other: Combined hyper- and hypoglycaemic clamp — During the entire clamp, participants will be monitored by ECG, pulse oximetry, and blood pressure and plasma glucose will be measured bedside every fifth minute. Additionally, patients with type 2 diabetes will be monitored by a loop recorder (LR) and a continuous glucose monitor (CGM). Comparison of LR and CGM recordings with the recordings obtained by ECG Holter monitor and blood sampling will be used for validation of the method used in Part 2 of the study. Blood samples will be drawn and analysed for changes in electrolytes, insulin, glucagon, catecholamines and cortisone. A cardiac haemodynamic evaluation will be performed by echocardiography at baseline, hyperglycaemia, and hypoglycaemia.
Device: Loop recorder (Reveal LINQ, Medtronic, Minneapolis, MN, USA) — Implantation of a loop-recorder
  Groups: Patients with type 2 diabetes
Device: Continuous glucose monitoring (iPro2, Medtronic, Minneapolis, MN, USA) — Monitoring with a continuous glucose monitor
  Groups: Patients with type 2 diabetes

SUMMARY:
Twenty-one patients with insulin-treated type 2 diabetes with diabetic complications will be recruited to Part 1 of the study, a three-hour combined hyper- and hypoglycaemic clamp, along with a control group of twenty-one individuals with normal glucose tolerance matched for age, gender, and body mass index. Patients with type 2 diabetes will be scheduled for a three-week run-in period with LR and CGM prior to participation in Part 1. Only patients with a well-functioning loop-recorder and who can comply with CGM will be included. Patients with type 2 diabetes will continue in part 2 of the study, a one year observational study employing CGM and LR and clinical examination after 1, 3, 6, 9, and 12 months and an extended observation period of 2 years employing LR and clinical examination.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes

* Informed and written consent
* Type 2 diabetes diagnosed according to the criteria of the World Health Organization (WHO)
* Treatment with insulin
* Glycated haemoglobin A1c (HbA1c) ≤58 mmol/mol
* One or more clinical relevant complications to diabetes defined as: peripheral neuropathy with vibration perception threshold of > 25 volt determined by biothesiometry, moderate to severe retinopathy, nephropathy (creatinine >130 μmol/l and/or albuminuria), and/or macrovascular disease. Macrovascular disease is defined as coronary disease (stable angina pectoris or previous unstable angina pectoris or myocardial infarct), cerebrovascular disease (previous stroke or transitional cerebral ischaemia), and peripheral vascular disease (previous intermittent claudication or prior acute ischemia)
* Well-functioning LR during run-in period (acceptable readings judged by an arrhythmologist)
* Participation in the extended study

Healthy individuals

* HbA1c ≤42 mmol/mol
* Fasting plasma glucose ≤6.1 mmol/l

Exclusion Criteria:

Patients with type 2 diabetes

* Arrhythmia diagnosed prior to or at the time of inclusion
* Implantable cardioverter defibrillator (ICD) or pacemaker at the time of inclusion
* Severe heart failure (left ventricular ejection fraction <25%)
* Structural heart disease (Wolf-Parkinson-White syndrome, congenital heart disease, severe valve disease)
* Insulin naïve patients with type 2 diabetes
* Thyroid dysfunction (except for well-regulated eltroxine substituted myxoedema)
* Unable to comply with daily CGM during run-in period
* Anemia (male: hemoglobin < 8.0; female: hemoglobin < 7.0 mmol/l)

Healthy individuals

* Type 1 or type 2 diabetes
* Prediabetes (HbA1c >42 mmol/l and/or fasting plasma glucose >6.1 mmol/l)
* Family history of diabetes (type 1 og type 2 diabetes)
* Arrhythmia diagnosed prior to or at the time of inclusion
* ICD or pacemaker at the time of inclusion
* Severe heart failure (left ventricular ejection fraction <25%)
* Structural heart disease (Wolf-Parkinson-White syndrome, congenital heart disease, severe valve disease)
* Thyroid dysfunction (except for well-regulated eltroxine substituted myxoedema)
* Anemia (male: hemoglobin < 8.0; female: hemoglobin < 7.0 mmol/l)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patiens with insulin-treated type 2 diabetes with complications and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Part 1: Clinically relevant arrhythmias | 0-240 min during the combined hyper- and hypoglycaemic clamp
  Composite endpoint including atrial fibrillation, brady-arrhythmias and tachy-arrhythmias. Clinically relevant brady-arrhythmias are defined as sinus arrest for more than 3 seconds, frequency below 30 beats per minute (bpm), or high grade atrioventricular (AV) block including Mobitz Type II and third-degree AV block. Clinically relevant tachy-arrhythmias are defined as sustained ventricular tachycardia (duration >30 seconds), and non-sustained ventricular tachycardia.
Part 2: Prevalence of clinically relevant arrhythmias as defined above | Within 12 months
  Prevalence of clinically relevant arrhythmias as defined above
Part 2: Clinically relevant arrhythmias during hypoglycaemia compared to euglycaemia | Within 12 months
  Clinically relevant arrhythmias during hypoglycaemia compared to euglycaemia
Part 2: Difference in MAGE | Within 12 months
  Difference in mean amplitude of glycaemic excursions (MAGE) two hours preceding an arrhythmic event versus MAGE during non-event

SECONDARY OUTCOMES:
Part 1: Differences in mean corrected QT interval (QTc) | 0-240 min during the combined hyper- and hypoglycaemic clamp
  Differences in mean corrected QT interval (QTc) between patients with type 2 diabetes and matched normal glucose tolerant individuals during the combined hyper- and hypoglycaemic clamp
Part 1: Difference in counter regulatory hormonal response | 0-240 min during the combined hyper- and hypoglycaemic clamp
  Difference in counter regulatory hormonal response between patients with type 2 diabetes and matched normal glucose tolerant individuals during the combined hyper- and hypoglycaemic clamp
Part 1: Differences in haemodynamic regulation | 0-240 min during the combined hyper- and hypoglycaemic clamp
  Differences in haemodynamic regulation (measured by echocardiography) between patients with type 2 diabetes and matched normal glucose tolerant individuals during a combined hyper- and hypoglycaemic clamp
Part 2: Clinical relevant arrhythmias during low glucose variability compared to high glucose variability. | Within 12 months
  Clinical relevant arrhythmias during low glucose variability (LGV), defined as variations in plasma glucose below or equal to 5 mmol/l within two hours preceding an arrhythmic event, compared to high glucose variability (HGV), defined as variations in plasma glucose above 5 mmol/l within two hours preceding an arrhythmic event
Part 2: The relationship between cardiovascular disease at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV | Within 12 months
  The relationship between cardiovascular disease (heart failure and ischaemic heart disease) at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV
Part 2: The relationship between pharmacological treatment at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV | Within 12 months
  The relationship between pharmacological treatment at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV
Part 2: The relationship between diabetes complication status at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV | Within 12 months
  The relationship between diabetes complication status (neuropathy, nephropathy, retinopathy) at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV
Part 2: Correlation between prevalence and total duration of hypoglycaemia and risk of clinically relevant arrhythmias | Within 12 months
  Correlation between prevalence and total duration of hypoglycaemia and risk of clinically relevant arrhythmias
Part 2: Correlation between plasma glucose variation and risk of clinical relevant arrhythmias | Within 12 months
  Correlation between plasma glucose variation (variation in plasma glucose (Δ mmol/l) within two hours of the event) and risk of clinical relevant arrhythmias

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Andersen A, Bagger JI, Sorensen SK, Baldassarre MPA, Pedersen-Bjergaard U, Forman JL, Gislason G, Lindhardt TB, Knop FK, Vilsboll T. Associations of hypoglycemia, glycemic variability and risk of cardiac arrhythmias in insulin-treated patients with type 2 diabetes: a prospective, observational study. Cardiovasc Diabetol. 2021 Dec 24;20(1):241. doi: 10.1186/s12933-021-01425-0. PMID 34952579